CLINICAL TRIAL: NCT03903341
Title: The Role of the Upper Colliculus in the Idiopathic Blepharospasm : a Pilot Study in Functional MRI
Brief Title: The Role of the Upper Colliculus in the Idiopathic Blepharospasm
Acronym: COLL-BSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC17.399
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Blepharospasm, Benign Essential
Keywords: Superior colliculus; fMRI
MeSH Terms: conditions — Benign essential blepharospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- idiopathic blepharospasm (BSP) de novo (Other): bold signal in visual pathway
  Interventions: Other: fMRI
- Healthy subjects (Other): bold signal in visual pathway
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — bold signal in visual pathway

SUMMARY:
This pilot study aims at investigating the role of superior colliculus in patients with idiopathic blepharospasm (BSP) de novo, compared to healthy subjects.

DETAILED DESCRIPTION:
The objective of the study is to investigate the function of the superior colliculus (SC) related to visual stimulation by means of fMRI (functional magnetic resonance imaging) in patients with idiopathic BSP compared to healthy subjects. The hypothesis is that SC function is impaired in BSP (role of biomarker of SC).

ELIGIBILITY:
Inclusion Criteria:

* Non treated idiopathic blepharospasm
* Age: 30- 70 years

Exclusion Criteria:

* Under the following treatments: Botulin toxin, anticholinergic, benzodiazepines, baclofen, beta- and alpha-blockers collyrium
* No MRI Contraindication

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Visual pathways fMRI | In a five months period after inclusion
  To measure the bold signal in superior colliculus and lateral geniculate corpus

CONTACTS AND LOCATIONS:
Overall Officials: Sara Meoni, MD, PhD, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, Grenoble, France